CLINICAL TRIAL: NCT05160103
Title: 16-Week Randomized Split-Face Efficacy Study of Cosmetic Formulations in Photoaged Pigmented Skin Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Avon Products, Inc. (Industry)
Collaborators: University of Cape Town, Groote Schuur Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 001-2021
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Aging Problems; Pigmentation
Keywords: cosmetic; ethnic skin; anti-aging; pigmentation

STUDY DESIGN:
Intervention Model Description: Single site, randomized, seven treatments, split face, efficacy study
Who Masked: Participant, Investigator
Masking Description: Products Codes A-G
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cosmetic Formulations — Topical emulsions containing anti-aging ingredients

SUMMARY:
The objective of this study is to determine the efficacy of seven different formulations currently marketed and commercially available cosmetic products on skin tone evenness, post-inflammatory hyperpigmentation, and discrete pigmentation in females of Fitzpatrick skin types IV-VI.

DETAILED DESCRIPTION:
This is a single site, double-blind randomized, split face, efficacy study. All subjects will receive a cleanser, Day Cream/sunscreen, and two treatment products. The treatment products will be applied in a split face fashion including behind the ear.

Local volunteer subjects will be enrolled such that a total of eighty-four (84) subjects will complete the study; with 24 subjects completing in each treatment.

Each subject will receive a cleanser, Day Cream/sunscreen and two treatment products as per the randomization. Subjects will use the cleanser twice daily, Day Cream/sunscreen in the morning, and the treatment products as specified after cleansing in the evening, for a period of 16 weeks. Clinical assessments, non-invasive instrument measurements and photographs will be completed at baseline and weeks 4, 8, 12, and 16. Biopsies will be taken at baseline and Week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Be a female in general good health, based on medical history reported by the subject;
2. From thirty (30) to sixty-five (65) years of age, inclusive;
3. Fitzpatrick skin types IV, V or VI;
4. Have mild to moderate skin tone evenness (a score of 3-6);
5. Willing to avoid excessive solar or UV exposure including: minimizing direct sun exposure and avoiding tanning beds and sunless tanning products for the duration of the study;
6. Willing to cleanse the face and remove all facial and all eye make-up prior to (or upon arrival) every study visit;
7. Willing to use no other topical products on the face for the duration of the study except the assigned test product and the subject's regular brand(s) of non-medicated make-up products that do not contain salicylic acid, benzoyl peroxide, AHA's, retinol, or their analogs or derivatives;
8. Willing to refrain from using exfoliating products for the duration of the study;
9. Not make any changes to her usual skin care regimen while participating in this study, other than those required by the study protocol;
10. Willing and able to follow all study instructions and adhere to study restrictions;
11. Read and sign an IRB approved informed consent form after the nature of the study has been fully explained and all questions have been answered by site staff;
12. Female subjects determined to be of child-bearing potential must indicate that they are not pregnant and/or lactating, nor do they intend to become pregnant during their study participation;
13. Female subjects determined to be of child-bearing potential must agree to practice a medically acceptable form of birth control during the study;

Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include:

* Established use of hormonal methods of contraception (oral, injected, implanted, patch or vaginal ring)
* Barrier methods of contraception (condom or diaphragm)
* Intrauterine device or system (IUD/IUS)
* Surgical sterilization (vasectomy, hysterectomy, tubal occlusion, uterine ablation)
* Abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence is not an acceptable method of contraception

Exclusion Criteria:

1. Has participated in any other clinical facial use study within four (4) weeks from the start of the study;
2. Has received any type of skin treatment or procedure in the past 3 (3) months including: chemical peels, microdermabrasion, injection of collagen or other filler, Botox® injections, or any treatment involving heat, light, or RF energy;
3. Is currently under a physician's care for a medical problem that, in the opinion of the Investigator or his designee, could affect the subject's treatment response;
4. Is nursing, pregnant, or planning a pregnancy during the course of this study;
5. Has excessive facial hair, or scars which could interfere with study evaluation in the opinion of the Investigator;
6. Is taking any prescription or over-the-counter medication that, in the opinion of the Investigator or his designee, could affect the subject's treatment response;
7. Has any other condition that, in the opinion of the Investigator or his designee, could interfere with the subject's ability to use the treatment as instructed, alter treatment response, or affect their ability to complete the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identifying females
Enrollment: 84 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Skin Tone Unevenness | Every 4 weeks up to 16 weeks
  Using a 0-9 scale where 0= even tone and 9=severe blotchy hyperpigmentation. Subjects will be recruited with mild to moderate skin tone unevenness. The goal is to show improvements by dermatologist assessments and photography
Skin Firming | Every 4 weeks up to 16 weeks
  Using a non-invasive clinical instrument (Cutometer) skin elasticity will be measure of the facial cheek
Skin Moisture | Every 4 weeks up to 16 weeks
  Using a non-invasive clinical instrument (SkiCon) skin conductance will be measure of the facial cheek
Skin Oiliness | Every 4 weeks up to 16 weeks
  Using a non-invasive clinical instrument (Sebumeter) skin conductance will be measure of the facial cheek

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Bayat, PhD, Principal Investigator — Professor & Co-Director, University of Cape Town

IPD SHARING:
Plan to Share IPD: No